CLINICAL TRIAL: NCT02554305
Title: The Fusion Versus The Affinity Oxygenation Systems - A Prospective Randomized Trial In Patients Undergoing Coronary Artery Bypass Grafting (CABG)
Brief Title: The Fusion Versus The Affinity Oxygenation Systems
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Oz Shapira, DIRECTOR OF THE DEPARTMENT OF CARDIOTHORACIC SURGERY, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 0033-15-HMO
Record Dates: First submitted 2015-08-09; First posted 2015-09-18 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Complication of Coronary Artery Bypass Graft
Keywords: efficacy and safety of fusion Oxygenation System; isolated Coronary Artery Bypass Grafting; Bypass Grafting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fusion oxygenation system (Active Comparator): Fusion oxygenation machine will be used during the operation.
  Interventions: Device: fusion oxygenation system
- Affinity oxygenation system (Active Comparator): Affinity oxygenation machine will be used during the operation.
  Interventions: Device: Affinity oxygenation system
- Peripheral vascular procedure (No Intervention): No oxygenation machine will be used in this group
- percutaneous coronary intervention (No Intervention): No oxygenation machine will be used in this group

INTERVENTIONS:
Device: fusion oxygenation system — The fusion oxygenation system is a novel design of the pump oxygenator used in cardiopulmonary bypass, integrating multiple new engineering concepts that have altered its performance profile.
  Arms: Fusion oxygenation system
Device: Affinity oxygenation system — The affinity oxygenation system is the classical pump oxygenator used in cardiopulmonary bypass surgeries
  Arms: Affinity oxygenation system

SUMMARY:
This study compares between the clinical, hematological, inflammatory and neurological outcome of patients undergoing Coronary Artery Bypass Grafting (CABG) surgery in which different oxygenation systems will be used.

DETAILED DESCRIPTION:
In order to assess the efficacy and safety of fusion Oxygenation System in patients undergoing isolated CABG, a prospective one-to-one randomized trial comparing the fusion oxygenation to the currently used affinity oxygenation system will be conducted. Forty patients intending to undergo CABG will be divided into 2 groups according to the oxygenation system which will be used during surgery. Distribution into groups will be done randomly. Ten patients undergoing elective peripheral vascular surgical procedures under general anesthesia and 10 patients undergoing elective percutaneous coronary intervention will serve as control groups for the neurological outcomes. Clinical status, inflammatory and hematological response as well as Neurological outcome will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-75 years old) undergoing first-time, isolated CABG at the Hebrew University, Hadassah Medical Center, Jerusalem, Israel and the University Hospital of Angers, Angers, France.
* Patients undergoing elective peripheral vascular surgical procedures under general anesthesia
* Patients undergoing elective percutaneous coronary intervention will serve as control groups

Exclusion Criteria:

* Emergency operations
* Left ventricular ejection fraction less than 30%
* CABG with concomitant procedure
* Previous stroke or documented neurological disorder
* High grade (>70%) unilateral or bilateral carotid stenosis
* Contraindication to MRI testing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
major adverse events | Participants will be followed for 30 days following the surgery
  Number of major adverse events (including mortality) will be assessed

SECONDARY OUTCOMES:
Systemic inflammatory response | Participants will be followed 3 days following the surgery.
  Serum markers of inflammation will be measured at 4 time points: after induction of anesthesia, immediately after termination of cardiopulmonary bypass, 3 hours, and 3 days postoperatively. : heparinized arterial (intraoperatively) or venous (postoperatively) blood samples will be collected. Bio-assay of endothelial permeability will be also done. Within each group, the change overtime will be compared to baseline. Participants' number with abnormal laboratory values in each study group will be assessed and compared with the other groups.
Number of participants with abnormal laboratory values | Participants will be followed for 3 days following the surgery.
  Hemoglobin and hematocrit, Platelet number and activation and Thrombin activation will be measured. Within each group, the change overtime will be compared to baseline. Participants' number with abnormal laboratory values in each study group will be assessed and compared with the other groups.
Neurological outcomes-Functional magnetic resonance imaging (MRI) | Changes in brain activity pattern will be assessed at baseline and 4 weeks postoperatively .
  Changes in brain structure and patterns of neural activation in response to cognitive tasks will be assessed using structural and functional MRI and compared between the study groups.
Neurological outcomes-Transcranial Doppler (TCD) | Participants will be followed 3 days following the surgery.
  Changes in brain activity pattern before and after the surgery will be assessed and compared between the study groups.
Neurological outcomes- electroencephalogram (EEG) | Participants will be followed 3 days following the surgery.
  Changes in brain activity pattern before and after the surgery will be assessed and compared between the study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Oz Shapira, MD, Principal Investigator — Hadassah Medical Organization